CLINICAL TRIAL: NCT01476228
Title: EEG Objectification in Neuropsychiatry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0394-11-HMO-CTIL
Record Dates: First submitted 2011-08-22; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-08

CONDITIONS: Personality Disorder; Depression; Neurodegeneration; Alzheimer's Disease; Epilepsy
MeSH Terms: conditions — Personality Disorders; Depression; Nerve Degeneration; Alzheimer Disease; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group (Experimental): EEG recording
  Interventions: Device: EEG recording

INTERVENTIONS:
Device: EEG recording — EEG recording

SUMMARY:
The main objective of the study is to evaluate the use of EEG in the management and follow-up of neuropsychiatric disorders. Secondary objectives are therefore better understanding of the pathological activations in neural network during neuropsychiatric disorders, their clinical evolution and response to therapies.

DETAILED DESCRIPTION:
Patients are having EEG recordings as a routine part of their clinical evaluation and diagnosis. EEG recording is harmless, has no side effects, any radiation or any mechanical or electrical influence. It is of short duration and may be done in the EEG institute or the patient's room.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of the investigated neuropsychiatric disease

Exclusion Criteria:

* Other co-existing neuropsychiatric conditions
* Refusal to participate in the study

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
percentage of fitting (0-100%) of EEG pattern to a previously identified electrophysiological "key" | 1 year
  The study will decode an EEG-based "key" (or electrophysiological pattern) for specific effect (such as the use of anti-epileptic agent or a certain condition) by comparing EEG before and after the use of this agent. For each patient the statistical fitting of the recorded EEG to the key will be evaluated by percentage (0-100%), describing fitting of the individual patient's EEG to the identified key.

CONTACTS AND LOCATIONS:
Overall Officials: shahar arzy, MD PhD, Principal Investigator — HMO
Locations (1):
- HMO, Jerusalem, Israel

REFERENCES:
- [Result] Arzy S, Collette S, Wissmeyer M, Lazeyras F, Kaplan PW, Blanke O. Psychogenic amnesia and self-identity: a multimodal functional investigation. Eur J Neurol. 2011 Dec;18(12):1422-5. doi: 10.1111/j.1468-1331.2011.03423.x. Epub 2011 May 7. PMID 21554495
- [Result] Arzy S, Allali G, Brunet D, Michel CM, Kaplan PW, Seeck M. Antiepileptic drugs modify power of high EEG frequencies and their neural generators. Eur J Neurol. 2010 Oct;17(10):1308-12. doi: 10.1111/j.1468-1331.2010.03018.x. PMID 20402743